CLINICAL TRIAL: NCT00422175
Title: A First-in-Human Study for BAF312: A Two Parts, Single Center, Randomized, Double-Blind, Placebo-Controlled Ascending Single Dose Study to Explore the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Oral BAF312 in Healthy Volunteers
Brief Title: Single Dose Study to Assess the Safety, Tolerability, Concentration in Body and Effect of BAF312
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBAF312A2101
Record Dates: First submitted 2007-01-11; First posted 2007-01-15 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Healthy
Keywords: Safety, tolerability, pharmacokinetics, pharmacodynamics, oral, BAF312, healthy volunteers
MeSH Terms: interventions — siponimod

INTERVENTIONS:
Drug: BAF 312

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and effect of oral BAF312 on bodily functions as well as the body's absorption, distribution, metabolism, and excretion of BAF312 in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 18 to 55 years of age included, and in good health
* Female subjects must be either surgically sterilized at least 6 months prior to study participation or post-menopausal (no regular menstrual bleeding for at least 1 years)
* Female subjects test are required to have a negative result for a pregnancy test, not be lactating/breast feeding, and must either:
* Body mass index (BMI) must be within the range of 18 to 30 Kg/m2. Subjects must weigh at least 50 kg to participate in this study.
* Able to communicate with the investigator, to understand and comply with the requirements of the study
* Understand and sign the written informed consent firm

Exclusion Criteria:

* Smokers
* Subjects who received live vaccine 4 weeks prior to dosing.
* Use of any prescription drugs four weeks prior dosing, or over-the-counter (OTC) medication (vitamins, herbal supplements, dietary supplements) within two weeks prior to dosing. Acetaminophen is acceptable
* Participation in any clinical investigation within 4 weeks prior to dosing or longer if required by local regulations, and for any other limitation of participation based on local regulations.
* Donation or loss of 400 ml or more of blood within 8 weeks prior to first dosing, or longer if required by local regulation.
* Significant illness within two weeks prior to dosing.
* A past personal or close family medical history of clinically significant cardiac abnormalities
* History of Acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease) Clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis) Known hypersensitivity or severe adverse event to darifenacin or similar drugs Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize participation in the study Immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result Positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result. Drug or alcohol abuse

Additional protocol defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63
Dates: Start 2006-10; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
safety, tolerability, and pharmacokinetic profile
Maximum Tolerated Dose

SECONDARY OUTCOMES:
Lymphocyte counts and lymphocyte recovery period
Cardiac rate and rhythm
Pulmonary function

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigative site
Locations (1):
- Novartis, East Hanover, New Jersey, United States